CLINICAL TRIAL: NCT01290822
Title: Optimized Biventricular Pacing in Allograft Recipients
Brief Title: Optimized Biventricular Pacing Allograft Recipients
Acronym: BiBET
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual and anticipated loss of funding
Sponsor: Henry M. Spotnitz (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Henry M. Spotnitz, George H. Humphreys, II Professor of Surgery, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAC1492; 1R01HL080152-01A2 (NIH)
Record Dates: First submitted 2011-02-02; First posted 2011-02-07 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Dilated Cardiomyopathy; Ischemic Cardiomyopathy
Keywords: Biventricular pacing; Dilated Cardiomyopathy; Ischemic Cardiomyopathy; Congestive heart failure; Cardiac allograft; Cardiac surgery; AVD; VVD; LV pacing site; pacing optimization
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BiVP Pacing (Experimental): BIVP optimize AVD, VVD, and LVPS parameters and assess the effect on cardiac output.
  Interventions: Device: BiVP
- AAI Pacing (Active Comparator): Traditional atrial (AAI) pacing
  Interventions: Device: AAI Pacing

INTERVENTIONS:
Device: BiVP — Biventricular pacing
  Other Names: Biventricular Pacing
  Arms: BiVP Pacing
Device: AAI Pacing — Atrial pacing
  Other Names: Atrial Pacing
  Arms: AAI Pacing

SUMMARY:
This study tests optimization of biventricular pacing (BiVP) in patients with dilated cardiomyopathy (DCM) or ischemic cardiomyopathy (ICM) during cardiac transplantation in patients with advanced cardiac failure. It examines the effects of atrioventricular delay (AVD), interventricular delay (VVD or RLD), and left ventricular pacing site (LVPS) on cardiac output (CO). BiVP results are compared to traditional atrial (AAI) pacing at an identical heart rate.

DETAILED DESCRIPTION:
This study is designed to increase the benefit of biventricular pacing (BiVP), which is an established therapy for advanced heart failure. The investigators will test 6 left ventricular (LV) pacing sites and 16 timing sequences in the operating room just before cardiac transplant. Pacing will be implemented after patients have been anticoagulated and connected to the heart-lung machine. Pacing by previously implanted pacemakers will be suppressed. The investigators will measure cardiac output (CO) by aortic flow probe (AFP), left ventricular (LV) contractility by a combination of trans-septal pressure gradients, and simultaneous left ventricular pressure (LVP)and transesophageal echocardiography (TEE) during transient reduction of inflow of blood to the heart by vena caval occlusion. The goal is to prove that this optimization will increase the amount of blood pumped by the failing heart by 15% as compared with standard atrial (AAI) pacing. The testing protocol is 12.5 minutes in duration, and the entire protocol should be executable in 20 minutes. Care will not be altered otherwise. Results will improve management of the general population of patients with advanced heart failure while minimally increasing the risk to patients undergoing cardiac transplantation. Benefits of this study should include: improved patient selection for BiVP and a decrease in the presently recognized 30-40% incidence of BiVP nonresponders.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) heart failure class III/IV
* Left Ventricular Ejection Fraction (LVEF) <36%
* QRS >120 msec

Exclusion Criteria:

* Intracardiac shunts
* Sinus tachycardia >120 bpm
* Second or third degree heart block
* Previous cardiac surgery
* Mechanical circulatory assistance
* Atrial fibrillation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry M Spotnitz, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medial Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data could not be analyzed due to poor enrollment and lack of data. "Per Arm" information is not available for the 1 subject who completed the study. It is also not available for the rest of the subjects as they were withdrawn before being studied.
Groups:
- All Subjects in the Study: This includes all subjects in the study. "Per Arm" information is not available for the 1 subject who completed the study. It is also not available for the rest of the subjects as they were withdrawn before being studied.
Period: Overall Study
Arm/Group | All Subjects in the Study
Started | 12
Completed | 1
Not Completed | 11
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 10

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects in the Study
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Output
Description: The primary endpoint of this study compares cardiac output between AAI pacing and optimal BiVP for DCM and ICM groups separately.
Time Frame: 13 minutes of testing; performed before CPB for allograft receipt
Population: Results could not be analyzed due to poor enrollment and lack of data.
Groups:
- All Subjects in the Study: This includes all subjects in the study
Arm/Group | All Subjects in the Study
Number analyzed (Participants) | 0

2. Secondary Outcome: Atrial Latency
Time Frame: 13 minutes of testing; performed before CPB for allograft receipt
Population: Results could not be analyzed due to poor enrollment and lack of data.
Arm/Group | All Subjects in the Study
Number analyzed (Participants) | 0

3. Secondary Outcome: Interatrial Delay (Between Right Atrium and Left Atrium)
Description: Results could not be analyzed due to poor enrollment and lack of data.
Time Frame: 13 minutes of testing; performed before CPB for allograft receipt
Arm/Group | All Subjects in the Study
Number analyzed (Participants) | 0

4. Secondary Outcome: Peak LV dP/dt
Time Frame: 13 minutes of testing; performed before CPB for allograft receipt
Population: Results could not be analyzed due to poor enrollment and lack of data.
Arm/Group | All Subjects in the Study
Number analyzed (Participants) | 0

5. Secondary Outcome: Peak RV dP/dt
Time Frame: 13 minutes of testing; performed before CPB for allograft receipt
Population: Results could not be analyzed due to poor enrollment and lack of data.
Arm/Group | All Subjects in the Study
Number analyzed (Participants) | 0

6. Secondary Outcome: Interventricular Synchrony
Time Frame: 13 minutes of testing; performed before CPB for allograft receipt
Population: Results could not be analyzed due to poor enrollment and lack of data.
Arm/Group | All Subjects in the Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse Events are not available due to poor enrollment and lack of data.
Arm/Group | All Subjects in the Study
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes